CLINICAL TRIAL: NCT06035562
Title: Promoting Positive Emotional Functioning in Police and Military Populations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Kevin Barber, Principal Investigator, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS26055 (H2023:201)
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Anhedonia
MeSH Terms: conditions — Anhedonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PVSET (Experimental): Participants will receive a course of individual therapy through the Operational Stress Injury Clinic (OSIC) at Deer Lodge Centre. Therapy will consist of a validated treatment protocol known as Positive Valence System Enhancement Treatment for Anxiety and Depression (PVSET), which will consist of psychoeducation and positive activity interventions designed to increase positive emotions, cognitions, and behaviors. Therapy sessions will be facilitated by psychologists, licensed therapists (e.g., MSW, RPN), and/or graduate students in psychology under supervision at the OSIC. PVSET will consist of 6 sessions, each lasting one hour, and will be delivered either virtually or in-person at OSIC depending on patient preference.
  Interventions: Behavioral: PVSET

INTERVENTIONS:
Behavioral: PVSET — 6, one-hour sessions of individual therapy, consisting of Positive Valence System Enhancement Treatment for Anxiety and Depression (PVSET), which will consist of psychoeducation and positive activity interventions designed to increase positive emotions, cognitions, and behaviors.

SUMMARY:
This study will examine whether actively serving and veteran members of the Canadian Armed Forces (CAF) and Royal Canadian Mounted Police (RCMP) who complete a treatment targeting anhedonia symptoms and amplifying positive emotional processing: 1) experience significant symptom reductions in anxiety, trauma, and depressive symptoms; 2) report increased experience of positive emotions; 3) report improvements to broad functioning and quality of life; and 4) find the treatment to be highly tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Be an actively serving or veteran member of the CAF and RCMP;
* Have been referred to receive the treatment protocol at the OSIC at Deer Lodge Centre by a doctor or psychologist;
* Have previously participated in at least one evidence-based psychological treatment for depressive, anxiety, or trauma-and-stressor-related condition at OSIC but remain clinically symptomatic;
* Be able to speak, read, and write in English;
* Have no current psychosis, untreated bipolar disorder, or current suicidal ideation with plan and intent;
* Be on a stable medication regime and agree to not make changes for the duration of the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in depression symptoms | 6 weeks
  Change in depression symptoms based on the Patient Health Questionnaire-9 (PHQ-9). Scores on this scale range from 0-27, with higher scores indication more severe depression.
Change in anxiety symptoms | 6 weeks
  Change in anxiety symptoms based on the Overall Anxiety Severity and Impairment Scale (OASIS). Scores on this scale range from 0-20, with higher scores indication more severe anxiety.
Change in PTSD symptoms | 6 weeks
  Change in PTSD symptom severity based on the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5). Scores on this scale range from 0-80 with higher scores indicating greater symptom severity.

SECONDARY OUTCOMES:
Change in positive and negative affect | 6 weeks
  Change in positive and negative affect based on the Positive and Negative Affect Schedule (PANAS). Scores on the two subscales of this assessment range from 0-50, with higher scores on the positive affect subscale representing higher levels of positive affect, and lower scores on the negative affect subscale representing lower levels of negative affect.
Change in quality of life | 6 weeks
  Change in quality of life as measure by the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q-SF). Scores on this scale range from 0-70, and are converted to a percentage, with higher scores indicating greater life enjoyment and satisfaction.
Psychotherapy progress | 6 weeks
  Psychotherapy progress as measured by the Outcome Questionnaire 45 (OQ-45). A total score of all subscales ranges from 0 to 180, with higher scores indicating more severe distress and functional impairment.
Treatment acceptability | 6 weeks
  Acceptability of the treatment program based on responses to a Treatment Acceptability Questionnaire. Scores on this questionnaire range from 5-30 with higher scores indicating greater acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- Deer Lodge Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No